CLINICAL TRIAL: NCT05526976
Title: PERIoperative Holistic RIsk Factor SCreening in the Prevention of Persistent Pain
Acronym: PERISCOPEcare
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE002575
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pain, Chronic Post-Surgical
Keywords: Persistent postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PERISCOPE-care — Patients with planned elective surgery will be asked to complete the PERISCOP3E-Care questionnaire (modified-Althaus & Kalkman, DN4, HADS, Stait-trait, NRS, MPI, EQ-5D-5L) preoperative. One month and three months post op the patients will be contacted to check if they developed persistend postoperative pain and they will also complete questionnaires (DN4, HADS, Stait-trait, NRS, MPI and EQ-5D-5L).

SUMMARY:
Assessment and management for improved wellbeing after elective surgery (PERISCOP³E-Care) Diagnostic assessment tool evaluation and cut-off determination for participation in a transmural perioperative care program

DETAILED DESCRIPTION:
Adult patients (≥ 18y) who are planned to undergo an elective surgery at the University Hospital Antwerp, will be invited to participate. After signing the informed consent, they will be asked to complete questionnaires (PERISCOP3E-care; Kalkman & modified-Althaus, DN4, HADS, Stait-trait, NRS, MPIn EQ-5D-5L) that involve screening of the risk to develop persistend postoperative pain (PPSP).

The questionnaires will be completed via a survey link to the RedCap platform. Invites will be send out via the patient's e-mail.

Demograpic data and relevant medical history, surgery history, concomitant medication will be registered.

one month and three months post surgery the patients will be contacted to identicate if they developed PPSP. They will also be asked to complete quesionnaires (MPI, HADS, Stai-Trait, NRS, MPI, DN4). Based on this info, the cut-off value will be defined for the preoperative questionnaire. Analysis will be done for the sensitivity and specificity of the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adult patiënts (≥ 18 year)
* planned elective surgery @ University Hospital Antwerp

Exclusion Criteria:

* incapacitated
* cognitive dificit that makes it impossible to complete the questionnaires
* language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first 560 patients who will undergo an elective surgery and have a preop consultation with a pain physician.
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Cut-off determination | preoperative
  Cut-off score determination for Kalkman and modified-Althaus risk for the prevention of persistend pain post op. Determination of inclusion and exclusion in the transmural care path

SECONDARY OUTCOMES:
Postoperative pain | postoperative (day 0 or 1day post surgery)
  Determination with numeric rating schale, NRS (numeric rating scale). Values from 0-10 with 10 being the highest pain you can have.
Persistent postoperative pain | 1 month and 3months post surgery
  Determination of persistent postoperative pain via NRS (numeric rating scale). Values from 0-10 with 10 being the highest pain you can have.
The use of opioids | 1month and 3months post surgery
  Need for daily intake of opioids (started postoperative) after surgery
The patients well-being | preoperative, 1month and 3months post surgery
  Evaluation of the well-being measured with EQ-5D-5L questionnaire (5-level EQ-5D version). Each dimension has 5 levels of response. (Level 1); slight; moderate; severe; and extreme problems (Level 5). here are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Fear and Depression | preoperative, 1month and 3months post surgery
  Evaluate the core complaints of fear and depression (without physical complaints) using the HADS questionnaire. Seven questions related to fear and seven questions related to depression. Every question can be answered with 0-1-2-3. If the score for the questions with fear is >8, this will indicate a psychiatric condition. If the score for the questions related to depression >8, this will indicate a psychiatric condition.
State anxiety and fear predisposition | preoperative, 1month and 3months post surgery
  Evaluation of the state anxiety and fear disposition using the Stai-Trait questionnaire. The range of scoring goes from a minimum of 20 untill a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80)
Pain complaints | preoperative, 1month and 3months post surgery if the NRS ≥ 3
  The MPI questionnaire part 1 measures the impact of pain on an individual's life, quality of social support and general activity. Each item is rated on a 0-6 scale, and the scoreds for each subscale are calculated by adding the score for each item in that subscale, devided by the number of items that subscale to yeald a mean score.
Neuropatic pain | preoperative, 1month and 3months post surgery if the NRS ≥ 3
  Evaluation of the presence of neuropatic pain components using the DN4 quesionnaire. When the score ≥ 4, neuropatic pain is likely.

CONTACTS AND LOCATIONS:
Overall Officials: Davina Wildemeersch, Principal Investigator — Staff Member
Locations (2):
- Belgium (2):
  - UZA, Edegem, Antwerp
  - University Hospital Antwerp, Antwerp

REFERENCES:
- [Derived] Wildemeersch D, Wauters E, Roelant E, Verhaegen I, De Clerck GR, Dankerlui R, Saldien V, Hans GH. A Novel Presurgical Risk Prediction Model for Chronic Post-Surgical Pain in Adults Undergoing Surgical Procedures: Development and Internal Validation of the P4-Prevoque Questionnaire [PERISCOPE Trial]. J Pain Res. 2025 Jul 5;18:3415-3428. doi: 10.2147/JPR.S525692. eCollection 2025. PMID 40636548
- [Derived] Wildemeersch D, Meeus I, Wauters E, Vanlommel L, Roelant E, Dankerlui R, Saldien V, Vandervelde L, Verhaegen I, Hans GH. Evaluating the Predictive Value of a Short Preoperative Holistic Risk Factor Screening Questionnaire in Preventing Persistent Pain in Elective Adult Surgery: Study Protocol for a Prospective Observational Pragmatic Trial [PERISCOPE]. J Pain Res. 2023 Dec 13;16:4281-4287. doi: 10.2147/JPR.S439824. eCollection 2023. PMID 38107366